CLINICAL TRIAL: NCT05000385
Title: Association of Masticatory Efficiency With the Condition of the Stomatognathic System in Children
Brief Title: Masticatory Efficiency in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinical Hospital Center Rijeka (Other)
Responsible Party: Principal Investigator, Odri Cicvarić, DMD, Principal Investigator, Clinical Hospital Center Rijeka
Other Study IDs: 1111
Record Dates: First submitted 2021-07-22; First posted 2021-08-11 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Mastication Disorder
Keywords: Body Mass Index; Child; Mastication; Stomatognathic Diseases; Particle size
MeSH Terms: conditions — Stomatognathic Diseases | interventions — Body Mass Index

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy: healthy complete dentition
  Interventions: Other: Assesment of masticatory efficiency with optical scanning method; Diagnostic Test: body mass index
- Dental caries: complete dentition with bilateral dental caries (ICDAS 4,5 or 6)
  Interventions: Other: Assesment of masticatory efficiency with optical scanning method; Diagnostic Test: body mass index
- Occlusal contacts: occlusal contacts are lost bilaterally due to extraction, changing dentition or orthodontic anomalies; no dental caries
  Interventions: Other: Assesment of masticatory efficiency with optical scanning method; Diagnostic Test: body mass index
- Dentures: patients with dentures, no caries and/or missing occlusal contacts on remaining teeth
  Interventions: Other: Assesment of masticatory efficiency with optical scanning method; Diagnostic Test: body mass index

INTERVENTIONS:
Other: Assesment of masticatory efficiency with optical scanning method — Participants will chew a standardized silicone tablet controlled by the examiner for 20 masticatory strokes. By scanning the comminuted particles, data on each particle size will be obtained. Enhanced masticatory performance is presented by a decrease in the chewed particle areas and an increase in the number of chewed particles.
Diagnostic Test: body mass index — as an indication of nutritional status

SUMMARY:
This study aims to evaluate the association of masticatory efficiency with different conditions of the stomatognathic system (transitioning from primary to secondary dentition, dental caries, malocclusion, tooth loss, prosthodontic treatment) in the paediatric population. Also, to assess the correlation between masticatory efficiency and nutritional status. The study will be conducted on children between 3 and 14 years of age. Masticatory efficiency will be evaluated by the optical scanning method. Participants will chew a standardized silicone tablet controlled by the examiner for 20 masticatory strokes. By scanning the comminuted particles, data on each particle's size will be obtained. Enhanced masticatory performance is presented by a decrease in the chewed particle areas and an increase in the number of chewed particles.

ELIGIBILITY:
Inclusion Criteria:

* children of both genders aged 3 to 14, with:

  * full healthy dentition
  * bilateral dental caries stage 4,5 or 6 by ICDAS criteria
  * reduced number of occlusal contacts
  * dentures
* signed informed consent by participant's parents
* verbal consent of the children

Exclusion Criteria:

* uncooperative behavior
* symptoms of temporomandibular joint dysfunction
* parafunctional habits
* systemic disturbances that can impact mastication
* ingestion of medicines that could interfere directly or indirectly with muscular activity
* tooth anomalies of structure, number or form
* periodontal disease
* tooth mobility

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children of both genders aged 3 to 14, with: full healthy dentition, bilateral dental caries stage 4,5 or 6 by ICDAS criteria, reduced number of occlusal contacts, and dentures, that are coming to Department of Paediatric Dentistry of Dental Clinic of the Clinical Hospital Center Rijeka for examination and/or therapy.
Sampling Method: Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
level of masticatory efficiency in children | 2 years
  determining the masticator efficiency variable (mean area of chewed particles) with optical scanning method, data comparison between four groups
masticatory efficiency and body mass index | 2 years
  determining the correlation of the masticatory efficiency variable (mean area of chewed particles determined by the optical scanning method) with body mass index (weight and height will be combined to report BMI in kg/m^2)

SECONDARY OUTCOMES:
dental caries and masticatory efficiency | 2 years
  determining the correlation of the masticatory efficiency (mean area of chewed particles determined by the optical scanning method) with the number of dental caries
occlusal contact and masticatory efficiency | 2 years
  determining the correlation of the masticatory efficiency (mean area of chewed particles determined by the optical scanning method) with the number of lost occlusal contacts

CONTACTS AND LOCATIONS:
Overall Officials: Odri Cicvaric, DMD, Principal Investigator — Department of Paediatric Dentistry, Faculty of Dental Medicine of the University of Rijeka
Locations (2):
- Croatia (2):
  - Clinical Hospital Center Rijeka, Rijeka, Primorje-Gorski Kotar County
  - Faculty of Dental Medicine of the University of Rijeka, Rijeka, Primorje-Gorski Kotar County